CLINICAL TRIAL: NCT05727345
Title: Comparison of Shoulder Anterior Capsular Block and Interscalene Brachial Plexus Block for Shoulder Arthroscopy: A Preliminary Analysis
Brief Title: Shoulder Anterior Capsular Block and Interscalene Brachial Plexus Block for Shoulder Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 142-2022
Record Dates: First submitted 2023-01-11; First posted 2023-02-14 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-02

CONDITIONS: Shoulder Arthroscopy; Interscalene Brachial Plexus Block; Shoulder Anterior Capsular Block; Rotator Cuff Rupture
Keywords: Shoulder arthroscopy; Postoperative pain; Interscalene brachial plexus block; Shoulder anterior capsular block; Hemodynamic stability
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Once the investigator chose from the opaque envelopes which group the patient will be included, interscalene brachial plexus block will be applied for Group A and shoulder anterior capsular block will be applied for Group B. All other interventions will be standardized.
Who Masked: Participant, Outcomes Assessor
Masking Description: After surgery, all patients will be followed by the same orthopaedist who is blind to the patient groups. Also, the patients themselves cannot know their groups as well. Only the investigator opens the opaque closed envelope and the same anesthesiologist, the investigator will perform blocks and will be the only one knowing study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene (Active Comparator): Right after general anesthesia induction and patient intubation, the patient will be placed in the semi-sitting position. Following sterile skin preparation, an interscalene block will be performed by the same anaesthesiologist under ultrasound guidance with an in-plane posterior approach approximately between C6-C7 nerve roots through a 22-gauge 50-mm insulated stimulating needle (StimuPlex Nanoline, Braun). Neurostimulation with an initial current of 0,5 mA, pulse width of 100ms, and a frequency of 2 Hz will be used as protection for intraneural injection, once the needle tip is in proximity to the brachial plexus. 15 mL local anesthetic solution (0.375 % bupivacaine anesthetic solution of 10 mL and 2 % lidocaine anesthetic solution of 5 mL) will be observed to disperse within the interscalene space.
  Interventions: Procedure: Interscalene brachial plexus block
- SHAC (Experimental): Right after general anesthesia induction and patient intubation, the patient will be placed in the semi-sitting position with the arm in extension and abduction. Following sterile skin preparation, a SHAC block will be performed by the same anaesthesiologist under ultrasound guidance by visualization of the interfascial space between the deep lamina of the deltoid muscle fascia and the superficial lamina of the subscapularis fascia and glenohumeral pericapsular space. A 22-gauge 50-mm insulated stimulating needle (StimuPlex Nanoline, Braun) will be used to give 1-3 mL of 5% Dextrose for the correct location and then 15 mL local anesthetic solution will be divided into 7,5 mL (0.375 % bupivacaine 5 mL and 2 % lidocaine 2,5 mL) for each target points as interfascial space and pericapsular space.
  Interventions: Procedure: Shoulder anterior capsular block

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — Preoperative ultrasound-guided interscalene brachial plexus block application
  Arms: Interscalene
Procedure: Shoulder anterior capsular block — Preoperative ultrasound-guided shoulder anterior capsular(SHAC) block application
  Arms: SHAC

SUMMARY:
The aim of our study is to reveal a comparison between interscalene brachial plexus block and shoulder anterior capsular block with respect to their efficacy on pain relief during perioperative anesthetic management. As intraoperative hemodynamic stability is an important factor for surgeons to achieve better outcomes because of its effect on the quality of arthroscopic visualization for shoulder arthroplasty, the investigators will also observe the effects of this matter.

50 patients scheduled for elective surgery will be randomized by closed envelope method into two groups (n=20) receiving either interscalene brachial plexus block or shoulder anterior capsular block preoperatively. Each group receives standardized general anesthesia and perioperative pain management protocol. Data to be recorded are numeric rating scales, intraoperative and postoperative analgesic use, intraoperative hemodynamic parameters, and arthroscopic visualization score. Moreover, block performance time, motor block, and side effects or complications will be noted.

DETAILED DESCRIPTION:
Introduction: Pain management after shoulder arthroplasty continues to be challenging. Although interscalene brachial plexus block has been accepted to be the gold standard intervention to relieve pain and improve postoperative outcomes by effecting functional rehabilitation and recovery times, usually results in motor block and complications such as hemi-diaphragmatic paralysis are possible to encounter. For this reason, the research for novel techniques to alleviate these outcomes resumes on the anatomical point of view and ultrasonography guidance. Shoulder anterior capsular block is a recently described interfascial and pericapsular block and is shown to be effective in relieving shoulder pain without motor block or complications.

The aim of our study is to reveal a comparison between interscalene brachial plexus block and shoulder anterior capsular block with respect to their efficacy on pain relief during perioperative anesthetic management along with intraoperative hemodynamic stability, and their effect on the quality of arthroscopic visualization for shoulder arthroplasty.

Material method: Patients scheduled for arthroscopic rotator cuff repair after June 30, 2022, are eligible for this study after ethical board approval. Inclusion criteria are (1) patients aged between 18-90 years with American Society of Anaesthesiologists (ASA) Physical Status classification I to III, (2) diagnosed with rotator cuff rupture, and (3) admitted receiving arthroscopic cuff repair surgery. Written informed consent will be obtained from all participants.

Exclusion criteria are refusal to participate in the study, history of neurologic deficits or neuropathy affecting the brachial plexus; infection at the site of the block application; coagulopathy; pre-existing respiratory dysfunction; allergy to local anesthetics; uncooperative patients who cannot reliably answer to verbal pain evaluation.

All patients will receive standard general anesthesia under standard monitorization; induction with 0,03 mg/kg midazolam, 2 mg/kg propofol, 2 mcg/kg fentanyl, 0,6 mg /kg rocuronium followed by 2% MAC sevoflurane in an air-oxygen mixture for maintenance of anesthesia. Randomization is designed with concealed opaque envelope in a 1:1 ratio into 2 block groups (n= 20): interscalene brachial plexus block (Group A) and shoulder anterior capsular block (Group B). All blocks will be performed before surgical incision by a single experienced regional anaesthesiologist (B.Ç.) under ultrasound guidance with the same local anesthetic doses: 0.375 % bupivacaine anesthetic solution of 10 mL and 2 % lidocaine anesthetic solution of 5 mL. The duration of the block procedure will be recorded by the anesthesia technician. Then the investigator will apply dexamethasone 4 mg (IV) after each block and approximately 15 minutes later the patient will be ready for a surgical incision. Intraoperative hemodynamic values (heart rate, systolic, and mean arterial pressure) will be recorded by the same technician. The same analgesia protocol will be applied as an infusion of remifentanil (0.01 to 0.1 μg · kg-1 · min-1) if only needed to maintain the heart rate and mean blood pressure within 20% of pre-induction values and 1 gr paracetamol. At the end of the surgery, the surgeon who is blind to the groups will decide the arthroscopic visualization score.

After surgery, all patients will be followed by the same orthopaedist who is blind to the patient groups. Also, the patients themselves cannot know their groups as well. Pain will be evaluated both by a numeric rating scale (0-10) and verbal rating scale starting at the post-anesthesia care unit (PACU) and at time intervals 2-6-12-24-48th hours postoperatively. Patients with persistent pain scores higher than 4 of 10 will receive rescue analgesia with 1mg/kg (maximum daily dose, 4x1) tramadol and 1 gr (maximum daily dose, 4x1) paracetamol. The duration of motor blockade if any, the severity of rebound pain and the total amount of analgesic drug used during the postoperative follow-up of the patient will be recorded. Before discharge, patient satisfaction (1. Not at all satisfied, 2. Dissatisfied 3. Moderate 4. Satisfied 5. Very satisfied) will be evaluated and the presence of postoperative side effects and complications will be questioned.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with rotator cuff rupture and admitted to receiving arthroscopic cuff repair surgery
* American Society of Anaesthesiologists (ASA) Physical Status classification I to III
* Patients who will give informed consent to peripheral nerve blocks

Exclusion Criteria:

* Refusal to participate in the study
* History of neurologic deficits or neuropathy affecting the brachial plexus
* Infection at the site of the block application
* Coagulopathy
* Pre-existing respiratory dysfunction
* Allergy to local anesthetics
* Uncooperated patients who cannot reliably answer verbal pain evaluation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | 2 days
  Numeric rating scale (NRS) worst pain imaginable as 10 points to zero pain. Verbal rating scale (VRS): no pain; slight pain; moderate pain; severe pain; unbearable pain
Analgesic drug used | 2 days
  The total amount of analgesic drug used during the postoperative follow-up

SECONDARY OUTCOMES:
heart rate | Intraoperative
  heart rate value at the monitor
Arthroscopic visualization score | Intraoperative
  arthroscopic visualization score: Grade 1: excellent; Grade 2: good sometimes cautery needed; Grade 3: moderate; often required cautery and manipulation; Grade 4: bad image
blood pressure | Intraoperative
  systolic arterial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, MD, Principal Investigator — Haseki Training and Research Hospital Anesthesiology and Reanimation Department
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamak Altinpulluk E, Teles AS, Galluccio F, Simon DG, Olea MS, Salazar C, Fajardo Perez M. Pericapsular nerve group block for postoperative shoulder pain: A cadaveric radiological evaluation. J Clin Anesth. 2020 Dec;67:110058. doi: 10.1016/j.jclinane.2020.110058. Epub 2020 Sep 26. No abstract available. PMID 32987232
- [Background] Kang R, Jeong JS, Chin KJ, Yoo JC, Lee JH, Choi SJ, Gwak MS, Hahm TS, Ko JS. Superior Trunk Block Provides Noninferior Analgesia Compared with Interscalene Brachial Plexus Block in Arthroscopic Shoulder Surgery. Anesthesiology. 2019 Dec;131(6):1316-1326. doi: 10.1097/ALN.0000000000002919. PMID 31490292